CLINICAL TRIAL: NCT06666881
Title: (Health Promotion) Skeletal Muscle Mass Changes on Images for Prediction of Prognosis After Exercise Training in Head and Neck Cancer Patients
Brief Title: Skeletal Muscle Mass Changes on Images for Prediction of Prognosis After Exercise Training in HNSCC Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wang Shao Chung, PhD, Professor Attending Physicians, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202201325A3
Record Dates: First submitted 2024-10-15; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer; Skeletal Muscle
Keywords: exercise training; dual energy X-ray absorptiometry; sarcopenia; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Sarcopenia

STUDY DESIGN:
Intervention Model Description: This project can determine the baseline skeletal muscle mass of Head and Neck cancer patients and hopes to monitor its changes after exercise training through imaging tools and find the most suitable imaging modalities. To understand the role of systemic inflammatory markers in sarcopenia,exercise training and Head and Neck cancer cancer prognosis. This study hopes to serve as a basis and reference for clinical treatment selection, imaging follow up, interventional treatment or rehabilitation. The results of this research should benefit patients in Taiwan and abroad, and to promote the medical treatment and health of patients.
Who Masked: Participant
Masking Description: group random
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): No Intervention: Head and Neck patients after CCRT treatment. After CCRT treatment, participants keep follow the skeletal muscle mass evaluation
- experimental (Experimental): Experimental: Head and Neck patients after CCRT treatment with exercise training.
  After CCRT treatment 4-5 week, arrange participants do the exercise training for patient. Two to three times a week ,total 24-36 times. Participants keep follow the skeletal muscle mass evaluation.
  Interventions: Other: HIIT only; Other: HIIT & Record of physical activities at home.

INTERVENTIONS:
Other: HIIT only — After CCRT treatment 4-5 week, arrange participants do the HIIT exercise for two to three times a week and total 24-36 times.
  Arms: experimental
Other: HIIT & Record of physical activities at home. — After CCRT treatment 4-5 week, arrange participants do the HIIT exercise for two to three times in a week and total 24-36 times. And do the recording of physical activities at home.
  Arms: experimental

SUMMARY:
This project adopts a prospective study design. It is scheduled to enroll 60 participants diagnosed with Head and Neck cancer in this hospital, of which 30 are in the experimental group and 30 are in the control group. The purpose of this research is to analyze the skeletal muscle mass changes on images in Head and Neck cancer patients after exercise training and the association with systemic inflammatory markers. Investigators would like to know whether these images and biomarkers predict the prognosis of Head and Neck cancer. Subjects enrolled in the trial will receive 36 times of exercise training after concurrent chemoradiotherapy. Before and after the completion of exercise training, investigators will arrange (1) dual energy X-ray absorptiometry (DXA) to measure the whole-body skeletal muscle mass and appendicular skeletal muscle mass and (2) blood tests for markers of systemic inflammation. In addition to DXA, computed tomography (CT) is another image modality for skeletal muscle mass evaluation. Positron emission tomography - CT or whole-body CT for cancer staging are considered as baseline studies. The routine follow-up CT images are used to analyze the changes after exercise training. If magnetic resonance imaging is also performed during the follow-up period, images will also be collected and assessed as an alternative.If the experimental group can maintain or even improve skeletal muscle mass and can be reflected in blood tests and prognosis, the result may be able to apply on cancer treatment and disease followup.

DETAILED DESCRIPTION:
This project adopts a prospective study design. It is scheduled to enroll 60 patients diagnosed with Head and Neck cancer in this hospital, of which 30 are in the experimental group and 30 are in the control group. The purpose of this research is to analyze the skeletal muscle mass changes on images in Head and Neck cancer participants after exercise training and the association with systemic inflammatory markers. Investigators would like to know whether these images and biomarkers predict the prognosis of head and neck cancer. Subjects enrolled in the trial will receive 36 times of exercise training after concurrent chemoradiotherapy. Before and after the completion of exercise training, investigators will arrange (1) dual energy X-ray absorptiometry (DXA) to measure the whole-body skeletal muscle mass and appendicular skeletal muscle mass and (2) blood tests for markers of systemic inflammation. In addition to DXA, computed tomography (CT) is another image modality for skeletal muscle mass evaluation. Positron emission tomography - CT or whole-body CT for cancer staging are considered as baseline studies. The routine follow-up CT images are used to analyze the changes after exercise training. If magnetic resonance imaging is also performed during the follow-up period, images will also be collected and assessed as an alternative. If the experimental group can maintain or even improve skeletal muscle mass and can be reflected in blood tests and prognosis, the result may be able to apply on cancer treatment and disease follow-up.

This project can determine the baseline skeletal muscle mass of Head and Neck cancer patients and hope to monitor its changes after exercise training through imaging tools and find the most suitable imaging modalities. To understand the role of systemic inflammatory markers in sarcopenia, exercise training and oral cancer prognosis. This study hopes to serve as a basis and reference for clinical treatment selection, imaging follow up, interventional treatment or rehabilitation. The results of this research should benefit participants in Taiwan and abroad, and to promote the medical treatment and health of participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20
2. Pathology:Squamous cell carcinoma
3. Need CCRT treatment
4. ECOG PS<2
5. Agree with blood drawing, exercise training, and all the procedures in the trial.

Exclusion Criteria:

1. ECOG PS≥2
2. Participants with intolerance basic exercise training, or without CCRT treatment
3. Mental illness or any medical illness or concurrent illness that may be aggravated by exercise training or unmanageable
4. Any medical condition that unsuitable for exercise training
5. refure to do the trial procedures: exercise training, blood drawing and all the procedures in the trial.
6. can't get the data for the whole-body computed tomography

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
dual energy X-ray absorptiometry data | baseline,pre-iprocedure
  measure the whole-body skeletal muscle mass
dual energy X-ray absorptiometry data | 3 month, during procedure
  measure the whole-body skeletal muscle mass
dual energy X-ray absorptiometry data | 8 month, during procedure
  measure the whole-body skeletal muscle mass

SECONDARY OUTCOMES:
Cardiopulmnary Exercise Test | baseline,pre-iprocedure
  record the VO2% of participants by doing the exercise test to assess the cardiopulmnary funtion before and after excercise training
Cardiopulmnary Exercise Test | 3 month, during procedure
  record the VO2% of participants by doing the exercise test to assess the cardiopulmnary funtion before and after excercise training
Cardiopulmnary Exercise Test | 8 month, during procedure
  record the VO2% of participants by doing the exercise test to assess the cardiopulmnary funtion before and after excercise training

OTHER OUTCOMES:
computed tomography (CT) | baseline,pre-iprocedure
  check toumor condition and another image modality for skeletal muscle mass evaluation
computed tomography (CT) | 8 month, during procedure
  check toumor condition and another image modality for skeletal muscle mass evaluation
blood data-myostatin | 3 month, during procedure
  inflammatory markers
blood data-myostatin | 8 month, during procedure
  inflammatory markers
blood data-IL-10 | 3 month, during procedure
  inflammatory markers
blood data-IL-10 | 8 month, during procedure
  inflammatory markers
blood data-IL-1β | 3 month, during procedure
  inflammatory markers
blood data-IL-1β | 8 month, during procedure
  inflammatory markers
blood data-IL-15 | 3 month, during procedure
  inflammatory markers
blood data-IL-15 | 8 month, during procedure
  inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Chung Wang, Study Director — New Taipei City TuCheng Hospital
Locations (1):
- New Taipei City TuCheng Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tieland M, Trouwborst I, Clark BC. Skeletal muscle performance and ageing. J Cachexia Sarcopenia Muscle. 2018 Feb;9(1):3-19. doi: 10.1002/jcsm.12238. Epub 2017 Nov 19. PMID 29151281